CLINICAL TRIAL: NCT04717973
Title: Comparison of Post-Operative Nutritional Deficiency Between Laparoscopic Sleeve Gastrectomy Versus Laparoscopic Gastric Bypass
Brief Title: Nutritional Deficiency After Bariatric Surgeries
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Farida Sami Abdou, assisstant lecturer of family medicine, Sohag University
Other Study IDs: Soh-Med-21-01-08
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Nutritional Deficiency
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients undergo sleeve gasterectomy
  Interventions: Diagnostic Test: laboratory testing of CBC, serum ferritin, and vitamin B 12
- patients undergo gasteric bypass
  Interventions: Diagnostic Test: laboratory testing of CBC, serum ferritin, and vitamin B 12

INTERVENTIONS:
Diagnostic Test: laboratory testing of CBC, serum ferritin, and vitamin B 12 — laboratory testing of CBC, serum ferritin, and vitamin B 12, vitamin D and ionized serum calcium after the 1st month, 3rd month, 6th month, and then after one year postoperative.
  The pre-operative and post-operative measures will be compared in patients who will be subjected to Laparoscopic Sleeve Gastrectomy versus Laparoscopic Gastric Bypass.
  Other Names: vitamin D and ionized serum calcium

SUMMARY:
comparing micro-nutrient deficiencies in postoperative morbid obese patients who will be undergoing gastric bypass and sleeve gastrectomy with regards to vit B 12, vitamin D,iron studies and calcium .

DETAILED DESCRIPTION:
The General surgery department will be reviewed for a period of six months duration. All patients who admitted to the department and subjected to laparoscopic GP and SG during the study period will be included in the study after securing an informed consent; both written and verbal consent approved by the Sohag Ethics Committee will be taken from all patients included in the study.

Patients will be followed for one year by laboratory testing of CBC, serum ferritin, and vitamin B 12, vitamin D and ionized serum calcium after the 1st month, 3rd month, 6th month, and then after one year postoperative.

The pre-operative and post-operative measures will be compared in patients who will be subjected to Laparoscopic Sleeve Gastrectomy versus Laparoscopic Gastric Bypass.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65.
2. BMI more than 40 and more than 30 with co morbidities
3. Both sexes with history of failed weight loss attempts in the past for two years and good motivation for surgery.

Exclusion Criteria:

1. Age less than 18, more than 65.
2. Revisional bariatric surgery.
3. Previous gastric surgery
4. Patients with endocrinal disturbance except hypothyroidism and DM
5. Psychological disturbed patients
6. Females during pregnancy

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The General surgery department will be reviewed for a period of six months duration. All patients who admitted to the department and subjected to laparoscopic GP and SG during the study period will be included in the study after securing an informedconsent; both written and verbal consent approved by the Sohag Ethics Committee will be taken from all patients included in the study postoperative.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
the degree of nutritional deficiency after gasteric bypass and sleeve gasterectomy 3 months postoperative | From Jan 2021 to april 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Farida sami abdou, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No